CLINICAL TRIAL: NCT01482208
Title: Study of Ultrasonic Hydration Monitor for Neonatology and Pediatric Children and Infants and/or Children up to Age 3 Years Old With Diarrhea
Brief Title: Clinical Evaluation of Ultrasonic Hydration Monitor for Infants
Acronym: IHM-01
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IHM-01; Gates Foundation (Other: Bill and Melinda Gates Foundation Round 6)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Diarrhea; Dehydration
Keywords: Dehydration; Hydration; Muscle composition; Diarrhea; Pediatrics; Neonatology; Ultrasound
MeSH Terms: conditions — Diarrhea; Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study will verify ability of infant Hydration Monitor (IHM) to assess changes of hydration status in newborns and infants by means of ultrasound velocity measurements through muscle tissues. Changes of tissue hydration will be followed during first days of life in newborns and in acute diarrhea in small children during re-hydration therapy. Weighting and clinical dehydration symptoms will be used as controls.

ELIGIBILITY:
Inclusion Criteria:

* Newborns from 1 to 7 days old,
* Health infants from 1 month to 3 years old,
* Any ethnicity,
* Male or female,
* Infants with diarrhea,
* Acute gastroenteritis,
* Diarrhea and/or vomiting,
* Suspected dehydration

Exclusion Criteria:

* Congenital heart disease,
* Renal failure,
* Chronic liver disease,
* Chronic lung disease,
* Inflammatory bowel disease,
* Immune deficiency,
* Severe malnutrition,
* Any external damage to skin of leg,
* Infants and Children whose parents refuse permission to be included

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns from 1 to 7 days Small children from 1 month to 3 years old
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Assess the ability of IHM to measure changes of hydration status ni newborn and infants | 1 week to several months
  Infants and small children diagnosed with diarrhea or presenting to the hopsital with diseases known to cause dehydration are eligible

CONTACTS AND LOCATIONS:
Overall Officials: Dace Gardovska, Dr. Med., Principal Investigator — Head of Pediatrics, CCUH RSU
Locations (1):
- Children Clinical University Hospital (CCUH) of the Riga Stradinsh University (RSU), Riga, Latvia

REFERENCES:
- See also: Sponsor Link to Reference #9 — http://www.artannlabs.com/publications.html